CLINICAL TRIAL: NCT05502822
Title: High Definition Transcranial Alternating Current Stimulation (HD-tACS) for Post-stroke Aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-TES-Aphaisa
Record Dates: First submitted 2022-07-26; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Transcranial Alternating Current Stimulation; Post-stroke Aphasia; Functional Magnetic Resonance Imaging
Keywords: Transcranial Alternating Current Stimulation; Functional Magnetic Resonance Imaging; Post-stroke Aphasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): Stimulation electrodes were arranged in a 4 × 1 ring configuration at F1, F2, C1 ,C2 and FCz, with the central one delivering an alternating current 2 mA and the surrounding 4 electrodes delivering one-fourth of the central electrode's current in the opposite polarity. The average peak-to-peak stimulation intensity across participants was 2 mA for the 6-Hz tACS. Participants will receive real tACS once daily for two weeks.
  Interventions: Device: High definition transcranial alternating current stimulation
- sham stimulation (Sham Comparator): In the sham condition, 6-Hz tACS was delivered only during the ramp-up and ramp-down periods (30 s); no current was delivered during the 30-minute intervention. Participants will receive sham tDCS once daily for two weeks.
  Interventions: Device: sham high definition transcranial alternating current stimulation

INTERVENTIONS:
Device: High definition transcranial alternating current stimulation — tACS is described as a non-invasive form of brain stimulation that uses a low-intensity, alternating current applied directly to the head through scalp electrodes.
  Arms: real stimulation
Device: sham high definition transcranial alternating current stimulation — . In the sham condition, 6-Hz tACS was delivered only during the ramp-up and ramp-down periods (30 s); no current was delivered during the 30-minute intervention.
  Arms: sham stimulation

SUMMARY:
To investigate the intervention effect of high definition transcranial alternating current stimulation(HD-tACS) in chronic post-stroke aphasia and its underlying neural mechanism by MRI.

DETAILED DESCRIPTION:
Aphasia is one of the most frequent cognitive deficits in poststroke survivor. More than 20% of stroke patients suffered from language impairment. The recovery of language dysfunction after stroke is highly variable. Some patients recover spontaneously in the early phases of stroke, but about two thirds of patients never fully restore language ability. The purpose of this study was to explore the intervention effect of high definition transcranial alternating current stimulation in chronic post-stroke aphasia.

40 patients with language disorder diagnosed by the Aphasia Battery of Chinese (ABC) were recruited from the first affiliated Hospital of Anhui Medical University. All participants underwent a structured interview and routine laboratory examination before and after receiving HD-tACS. After meeting the inclusion criteria and obtaining informed consent, each participant will complete the clinical evaluation, functional magnetic resonance imaging (fMRI) and HD-tACS treatment conducted by trained researchers at the Neuropsychological Synergetic Innovation Center of Anhui Medical University.

All the participants were randomized (1:1) to receive "real" or "sham" treatment protocol. Stimulation electrodes were arranged in a 4 × 1 ring configuration at F1, F2, C1 ,C2 and FCz, with the central one delivering an alternating current 2 mA and the surrounding 4 electrodes delivering one-fourth of the central electrode's current in the opposite polarity. The average peak-to-peak stimulation intensity across participants was 2 mA for the 6-Hz tACS. In the sham condition, 6-Hz tACS was delivered only during the ramp-up and ramp-down periods (30 s); no current was delivered during the 30-minute intervention. The tACS stimulation lasted 30 minutes, a duration that is common in cognitive neuroscience research. During the tACS, participants sat comfortably in front of a screen, training the speech and comprehension functions to follow a speech therapist.

Before and after the HD-tACS treatment, the patients had receiving a battery measure of neuropsychological tests and Magnetic resonance imaging scan in multimodalities. Neuropsychological assessment included ABC, VFT, Token, MMSE, MoCA, HAMD, HAMA, ADL. Multimodal fMRI includes 3D-T1, rs-fMRI, DTI and ASL.

Neuropsychological evaluation and magnetic resonance imaging data were obtained again 24 hours after the last treatment. The symptoms of the patients were followed up one month after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* aphasia diagnosed by the ABC.
* 18-75 years old.
* native Chinese speaker.
* right-handed.
* post onset of stroke ≥6months.

Exclusion Criteria:

* mental illness .
* severe dysarthria.
* a history of head injury or surgery.
* alcohol or substance abuse.
* cerebral tumor or abscess.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
language function | baseline and immediately after intervention
  Language deficit was assessed by the same professional language therapist using the Aphasia Battery of Chinese (ABC). The multidimensional test contains four subtypes, including spontaneous speech (semi-standardized interview, assessment of the fluency, and information of speech; total score 20 points), auditory comprehension (yes or no question, auditory picture matching task, and verbal instruction; total score 230 points), repetition (words and sentences; total score 100 points), and naming (simple objects, colors, pictures, and situations; total score 80 points). The combined score is used to calculate an aphasia quotient (AQ) reflecting the overall severity of language impairment. Patients with AQ below 93.8 points were considered as aphasic.
resting-state functional connectivity | baseline and immediately after intervention
  the change of resting-state functional connectivity strength between stimulated target and the whole brain areas will be measured by functional MRI.

SECONDARY OUTCOMES:
comprehension function | baseline and immediately after intervention
  the change of comprehension dysfunction will be assessed by Token. Token is composed of six parts. Token scale scores range from 0 to 36 points. Lower scores indicate more severe comprehension dysfunction.
MMSE(Mini Mental State Examination) | baseline and immediately after intervention
  The full name of MMSE is mini-mental state examination, and the scale consists of 30 subject, include the following seven aspects: time orientation, place orientation,immediate memory,attention and calculation,delay memory,language, visual space.One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answe he/she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Xie, Study Chair — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, China